CLINICAL TRIAL: NCT00010946
Title: Acupuncture Safety/Efficacy in Knee Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Masking: Single | Purpose: Treatment
Other Study IDs: U01 AT000171-01M; 1U01AT000171-01 (NIH); NCT00009490 (obsolete NCT alias)
Record Dates: First submitted 2001-02-02; First posted 2001-02-05 (Estimated); Last update posted 2008-03-07 (Estimated); Status verified 2008-03

CONDITIONS: Osteoarthritis, Knee
Keywords: acupuncture; osteoarthritis; elderly
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Acupuncture Therapy

INTERVENTIONS:
Procedure: Acupuncture

SUMMARY:
The goal of this research is to determine the efficacy and safety of Traditional Chinese Acupuncture (TCA) in patients with osteoarthritis of the knee. A three arm randomized controlled trial (RCT) using sham TCA, true TCA, and an education/attention comparison group with a total sample of 525 is proposed. Primary hypothesis to be tested is that patients randomized to true TCA will have significantly more improvement in pain and function as measured by the Womac Pain & Function Scales and patient global assessments than patients randomized to the sham acupuncture and education/attention control groups.

Secondary aims of the study are to 1) determine if improvement with TCA differs between patients below age 65 vs. those aged 65 and above, 2) to determine if improvement with TCA differs by racial/ethnic group (ie., Caucasian, Black, Hispanic), and 3) to determine if improvement with TCA differs by stage of radiographic severity of knee OA at baseline (KL grade 2, 3 or 4)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of osteoarthritis of the knee (fulfilling ACR criteria) for at least 6 months duration
* At least moderate pain in the knee for most days in the last month
* Must be taking analgesic or nonsteroidal anti-inflammatory agents for control of pain
* Documented radiographic changes of osteoarthritis (Kellgren-Lawrence grade>2) at the time of rheumatological screening
* Signed informed consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-09; Study Completion 2003-08

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Brian Berman, Principal Investigator — University of Maryland/Complementary Medicine Program
Locations (3):
- United States (3):
  - Kernan Hospital Mansion, Baltimore, Maryland
  - Catonsville Clinic, Catonsville, Maryland
  - Hospital for Special Surgery, New York, New York

REFERENCES:
- [Background] Berman BM, Singh BB, Lao L, Langenberg P, Li H, Hadhazy V, Bareta J, Hochberg M. A randomized trial of acupuncture as an adjunctive therapy in osteoarthritis of the knee. Rheumatology (Oxford). 1999 Apr;38(4):346-54. doi: 10.1093/rheumatology/38.4.346. PMID 10378713
- [Background] Berman BM, Lao L, Greene M, Anderson RW, Wong RH, Langenberg P, Hochberg MC. Efficacy of traditional Chinese acupuncture in the treatment of symptomatic knee osteoarthritis: a pilot study. Osteoarthritis Cartilage. 1995 Jun;3(2):139-42. doi: 10.1016/s1063-4584(05)80046-9. No abstract available. PMID 7584319